CLINICAL TRIAL: NCT01450618
Title: Comparative Tolerability of Protease Inhibitors and the Associated Impact on Persistence, Healthcare Utilization, and Healthcare Costs
Brief Title: Comparative Tolerability of Protease Inhibitors
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI424-435
Record Dates: First submitted 2011-09-21; First posted 2011-10-12 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Atazanavir: HIV patients on antiretroviral therapy using Atazanavir
- Darunavir: HIV patients on antiretroviral therapy using Darunavir
- Fosamprenavir: HIV patients on antiretroviral therapy using Fosamprenavir
- Lopinavir: HIV patients on antiretroviral therapy using Lopinavir

SUMMARY:
This study will be a retrospective observational study assessing identifiable tolerability problems in terms of their comparative incidence among Human Immunodeficiency Virus (HIV) patients treated with cART regimens including one of four different protease inhibitors [Atazanavir sulfate (ATV), Darunavir (DRV), Fosamprenavir (FPV), or Lopinavir (LPV)] and the impact of these identifiable tolerability problems on PI persistence, healthcare utilization, and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Initiated treatment with a Protease inhibitor (PI)-based Combination antiretroviral therapy (cART) regimen
* Between 18-64 years of age on the index date
* At least 6 months of continuous enrollment and pharmacy benefits prior to the index date
* At least 6 months of continuous enrollment and pharmacy benefits following the index date
* At least 1 medical claim during the 6-month follow-up period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Employees and dependents with employer-based health insurance coverage
Sampling Method: Non-Probability Sample
Enrollment: 26000 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Percent of patients.with new onset GI symptoms after initiating an ATV, DRV, FPV, or LPV containing combination antiretroviral therapy (cART) regimen | 6 months

SECONDARY OUTCOMES:
Percent of patients with new onset lipid abnormalities or new onset jaundice (separately) after initiating an ATV, DRV, FPV, or LPV containing combination antiretroviral therapy (cART) regimen | 6 months
Healthcare utilization | 6 months
Healthcare costs | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm